CLINICAL TRIAL: NCT06920277
Title: Data Collection for the Development of Artificial Intelligence (AI) Software to Support Ultrasound-Guided Regional Anesthesia Procedures
Brief Title: Ultrasound Image Collection for the Development of an AI Software
Status: Completed | Type: Observational
Sponsor: Smart Alfa Teknoloji San. ve Tic. A.S. (Industry)
Responsible Party: Sponsor
Other Study IDs: NRV-001-04
Record Dates: First submitted 2025-03-25; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Ultrasound Scan
Keywords: Data collection; Artificial Intelligence; Regional Anesthesia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- U.S. population
  Interventions: Device: Ultrasound scans

INTERVENTIONS:
Device: Ultrasound scans — 10 seconds scanning for one block region

SUMMARY:
This study is designed to collect ultrasound images from healthy volunteers in the U.S.

DETAILED DESCRIPTION:
The goal of this study is to create an ultrasound image dataset of healthy volunteers from the U.S. population. This dataset will be used for development of an AI software which will assist anesthesiologists in detection of key anatomical structures on the ultrasound image for peripheral nerve block applications. These blocks are:

* Interscalene Brachial Plexus
* Supraclavicular Brachial Plexus
* Infraclavicular Brachial Plexus
* Cervical Plexus
* Axillary Brachial Plexus
* PECS I & II
* Transversus Abdominis Plane (TAP)
* Rectus Sheath
* Femoral Nerve
* Adductor Canal
* Popliteal Sciatic
* Erector Spinae Plane (ESP)

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* At least 18 years of age and older
* Stated willingness to comply with all study procedures and availability for the duration of the study
* In good general health

Exclusion Criteria:

* Pregnancy
* Inability to lie to flat
* Any complaint or anatomical deformity on the regions to be scanned

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: volunteers from the U.S. population
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2024-10-29 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Number of ultrasound scan recordings relevant to peripheral nerve blocks collected | Day 1, 2 and 3
  Ultrasound scans will be collected and reviewed for quality and completeness. The outcome will be the number of ultrasound recordings that meet predefined criteria for image quality; correct anatomical region and clear visualization to support AI development.

CONTACTS AND LOCATIONS:
Overall Officials: Senanur Samur Duysal, Principal Investigator — Smart Alfa Teknoloji San. ve Tic. A.S.
Locations (1):
- Conference Room at Doubletree by Hilton Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No